CLINICAL TRIAL: NCT02348125
Title: Does Clinical Treatment of Mitochondrial Dysfunction Impact Autism Spectrum Disorder (ASD)?
Acronym: MitoASD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DrexelMitoApp
Record Dates: First submitted 2014-12-22; First posted 2015-01-28 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorders; Mitochondrial Diseases
MeSH Terms: conditions — Autism Spectrum Disorder; Mitochondrial Diseases | interventions — Carnitine; Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mitochondrial Cocktail (Experimental): The precise content of the Mitochondrial Cocktail will be:
  * ubiquinol (liquid form, 150 mg/kg subject weight/day
  * carnitine, 50 mg/kg subject weight/day
  * alpha-lipoic acid, 100 mg/ day
  Interventions: Drug: Mitochondrial Cocktail

INTERVENTIONS:
Drug: Mitochondrial Cocktail
  Other Names: Ubiqinol; Levocarnitine; Alpha Lipoic Acid

SUMMARY:
In this study, 50 children between 3 and 12 years old with formally diagnosed autistic spectrum disorders (ASD) and also having significant mitochondrial dysfunction will be treated for a 3 month period with the Mitochondrial Cocktail, a combination of specific nutritional supplements and metabolite intermediates (including anti-oxidants) and bio-energy substrates. A series of neurological and psychological evaluations will be conducted by trained evaluators/clinicians to evaluate both the severity and the clinical presentation of the ASD/mitochondrial dysfunction with each subject at baseline prior to treatment, after the 3 month treatment and again at 6 months, after another 3 month non-treatment period. In addition, laboratory investigations will be conducted at the same time-points to assess the mitochondrial dysfunction and cellular biomarkers thought to be associated with autistic and mitochondrial disorders. These investigations will include the analysis of samples of blood and cheek/buccal swabs collected from each child to assess select biochemical markers of ASD. The Mitochondrial Cocktail treatment will be administered at home once a day continuously for a total of 3 months. All the children in the study will be treated with the same Mitochondrial Cocktail (an open label study).

DETAILED DESCRIPTION:
In this study, 50 children between 3 and 12 years old with formally diagnosed autistic spectrum disorders (ASD) and also having significant mitochondrial dysfunction will be treated for a 3 month period with the Mitochondrial Cocktail, a combination of specific nutritional supplements and metabolite intermediates (including anti-oxidants) and bio-energy substrates. The Mitochondrial Cocktail is presently widely used as the standard of care for clinically treating mitochondrial dysfunction.

The precise content of the Mitochondrial Cocktail will be:

* ubiquinol (liquid form, 150 mg/kg subject weight/day
* carnitine, 50 mg/kg subject weight/day
* alpha-lipoic acid, 100 mg/ day.

A series of neurological and psychological evaluations will be conducted by trained evaluators/clinicians to evaluate both the severity and the clinical presentation of the ASD/mitochondrial dysfunction with each subject at baseline prior to treatment, after the 3 month treatment and again at 6 months, after another 3 month non-treatment period. In addition, laboratory investigations will be conducted at the same time-points to assess the mitochondrial dysfunction and cellular biomarkers thought to be associated with autistic and mitochondrial disorders. These investigations will include the analysis of samples of blood and cheek/buccal swabs collected from each child to assess select biochemical markers of ASD. The Mitochondrial Cocktail treatment will be administered at home preferably in the morning once a day continuously for a total of 3 months. All the children in the study will be treated with the same Mitochondrial Cocktail (an open label study). . Safety will be also evaluated based on the occurrence of adverse events either reported spontaneously by the subject and/or caregiver or observed by the investigator(s).

ELIGIBILITY:
Inclusion Criteria:

1. Subject/legal representative is considered reliable and capable of adhering to the protocol (e.g., able to understand and complete diaries), visit schedule, and medication intake according to the judgment of the investigator.

   .
2. Subject has a formal diagnosis of autistic spectrum disorders (ASD). the ASD diagnosis will satisfy the DSM- V criteria for ASD, and will be broad-spectrum including both severe and milder cases.
3. All subjects will have either suspected mitochondrial dysfunction as assessed by clinical evaluation, mitochondrial dysfunction as defined by the presence of significant abnormalities in their buccal mitochondrial respiratory complex activities (i.e., with either respiratory complex I or complex IV deficiencies) or have significantly aberrant specific activity ratios. Subjects with significant deficiencies in either muscle or skin fibroblast respiratory activities will also be included in those cases if buccal mitochondrial respiratory enzyme activity testing has not been performed.

Exclusion Criteria:

1. Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study.
2. Subject has a medical condition that could be expected in the opinion of the investigator to interfere with drug absorption, distribution, metabolism, or excretion.
3. Subject is on a ketogenic or other specialized diet. If the subject was on a specialized diet in the past, they must be off the diet for ≥2 months prior to the Baseline Period.
4. Subject has an acute or sub-acutely progressive central nervous system disease.
5. Subject has major brain deformation or severe cognitive dysfunction.
6. Subjects with epilepsy needing to take anti-seizure medications will be excluded.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in features of Autistic behavior phenotype assessed using the Social Responsiveness Scale (SRS) | Baseline (0), 3 and 6 months
Change in Executive Function assessed using the Behavior Rating Inventory of Executive Function (BRIEF) | Baseline (0), 3 and 6 months

SECONDARY OUTCOMES:
Changes in mitochondrial enzyme specific activities biochemically evaluated using buccal swab analysis | Baseline (0), 3 and 6 months
Change in buccal oxidative stress markers and mitochondrial DNA (mtDNA) damage | Baseline (0), 3 and 6 months
  In buccal extracts, aconitase activity levels and mtDNA levels and integrity will be quantitatively evaluated at 0,3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Goldenthal, PhD, Study Director — Drexel University College of Medicine
Locations (1):
- St. Christopher's Hospital for Children, Philadelphia, Pennsylvania, United States